CLINICAL TRIAL: NCT07113158
Title: Effect of Aspirin and Folic Acid for Sudden Sensorineural Hearing Loss
Acronym: SERORL
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APHP230836; 2024-513710-35 (EudraCT Number)
Record Dates: First submitted 2024-10-28; First posted 2025-08-08 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Sudden Sensorineural Hearing Loss
Keywords: SSNHL; sudden sensorineural hearing loss; sudden hearing loss; aspirin; acid folic
MeSH Terms: conditions — Hearing Loss, Sudden | interventions — Aspirin; Folic Acid

STUDY DESIGN:
Intervention Model Description: This is a national phase III, clinical study, multicenter, comparative, randomized on 2 parallel groups, with one group control, of superiority, double blind for the patients, the investigators and the study site staff. Participants distributed between groups at a ratio of (1: 1).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational medicinal products (Experimental): Aspirin 100 mg/day and Acid Folic 5 mg/day + gold standard treatment (oral corticosteroid therapy 1 mg/kg +/- 3 trans-tympanic injections of dexamethasone)
  * Corticosteroid therapy 1mg/kg/day for 7 days
  * 3 trans-tympanic injections of corticosteroids if hearing loss persists at D15 Duration of treatment: 3 months
  Interventions: Drug: Aspirin + Acid folic
- Comparator treatment (Placebo Comparator): The Placebo Aspirin 100 mg/j + Placebo folic acid 5 mg/j + reference treatment (oral corticosteroid therapy 1mg/kg +/- 3 trans-tympanic injections of dexamethasone)
  * Corticosteroid therapy 1mg/kg/day for 7 days
  * 3 trans-tympanic injections of corticosteroids if hearing loss persists at D15 Duration of treatment: 3 months
  Interventions: Drug: Placebo Aspirin + Placebo Acid folic

INTERVENTIONS:
Drug: Aspirin + Acid folic — Aspirin 100 mg/day and Acid Folic 5 mg/day + gold standard treatment
  Arms: Investigational medicinal products
Drug: Placebo Aspirin + Placebo Acid folic — The Placebo Aspirin 100 mg/j + Placebo folic acid 5 mg/j + reference treatment
  Arms: Comparator treatment

SUMMARY:
The annual incidence of sudden sensorineural hearing loss (SSNHL) is 5 to 20 per 100 000 persons. The pathophysiology of SSNHL and acute vestibulo-cochlear syndromes (VCS) is unknown in more than 70% of cases.

Hypothesis : an inner ear microvascular disease represents the key element in the pathogenesis of SSNHL and acute VCS.

Plasma serotonin has among other tissular effect a vasospastic on microcirculation such as the inner ear microvascularisation. Increased plasma homocysteine has a deleterious effect on vascular endothelium. Inner ear microvascularisation sensitized by an increased homocysteine level and the vascular wall would vasoconstrict under serotonin stimulation inducing ischemia of the vestibular and/or cochlear organs.

DETAILED DESCRIPTION:
Sudden sensorineural hearing loss (SSNHL) is defined as sensorineural hearing loss of 30dB or greater over at least three contiguous audiometric frequencies occurring over 72 hr 9,10. SSNHL is a relatively common disorder in otologic and audiologic practices (1.5-1.7 per 100 new patients presenting in ENT practice. Most patients with sudden SSNHL have no identifiable cause for hearing loss and are classified as "idiopathic". Despite extensive research, the etiology and therapeutic management of SSNHL and acute VCS remain elusive. Regardless of the etiology, complete or partial recovery of hearing thresholds following SSNHL may not occur. Factors influencing hearing recovery include the age at onset of hearing loss, severity and frequencies affected, the presence of vertigo, and the delay of treatment. The incidence of SSNHL is 5-20 per 100, 000. The true incidence of SSNHL may be higher than these estimates because affected individuals who recover spontaneously do not present for medical care. Although individuals of all ages can be affected, the peak incidence is between the fifth and sixth decade of life. Men and women are equally affected. Nearly all cases of SSNHL are unilateral; less than 2% of patients have bilateral involvement and typically bilateral involvement is sequential. Accompanying symptoms include tinnitus (41% to 90%) and dizziness (29% to 56%) New vestibular function assessment now allows us to specify the vestibular damage associated with SSNHL. Until now, the association with dizziness was a poor prognostic factor for hearing. In a recent study in 2023, more than 60% of patients treated for SSNHL had associated vestibular damage even if they did not complain of vestibular symptoms. 20. Vestibular involvement has often been under-diagnosed and could be a way of targeting more precisely the pathophysiological mechanisms behind SSNHL. Vestibular and cochlear damage can be secondary to a pressure disorder of the endolymphatic system (endolymphatic atelectasis or endolymphatic hydrops) or to microvascular damage of cochlear and/or vestibular arteries (e.g. cochlear artery syndrome), but also to inflammatory damage of the labyrinth. 3D-Flair Endolymph magnetic resonance imaging highlighted the different mechanisms involved in deafness: endolymphatic hydrops or atelectasis, microvascular or inflammatory involvement the presence or absence of a rupture of the blood-labyrinth barrier. For all these disorders, increase serum homocysteine and plasma serotonin levels would be a predisposing factor, weakening the microvascularisation inner ear's vascular endothelium.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral SSNHL defined as a sudden hearing loss of 30dB or greater at least three contiguous audiometric frequencies (between 125hz and 8000Hz) occurring within a 72 hr period and for less than 15 days.
* Individuals affiliated to a social security regimen
* Individuals able to participate and to follow up during the study period

Exclusion Criteria:

* Contra-indications to Aspirin, contra-indications to oral corticosteroid therapy, contra-indications to dexamethasone, allergy to vitamin B9
* Evident cause of acute SSNHL including tumor of the ponto-cerebellous angle, infectious labyrinthitis, mechanical and acoustic trauma, malformation of the inner ear, neurological disorder.
* Patient already including in another clinical trial
* Person under legal protection (under guardianship or curatorship)
* Patients taking serotonin reuptake inhibitors
* Patients already taking aspirin or other anticoagulant or antiplatelet agent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Mean PTA (mean of the change of the hearing thresholds for the 3 most affected contiguous frequencies) at D15 as defined by the AAO-HNS | At Day 15
  Complete recovery with return to less than 10 dB HL of the unaffected ear, no recovery : anything below 10 dB. Partial recovery is between the two extremes.

SECONDARY OUTCOMES:
Maximal speech intelligibility (word recognition) score at D15, M3 and M6 | At day 15, 3 month, 6 month
Mean of pure tones defined as the mean PTA (mean of the change of the hearing thresholds for the 3 most affected contiguous frequencies) at M3 and M6 as defined by the AAO-HNS | At month 3, month 6
  Complete recovery with return to less than 10 dB HL of the unaffected ear, no recovery : anything below 10 dB. Partial recovery is between the two extremes.
Quality of life will be evaluated with THI and DHI questionnaire at D15, M3 and M6 | At day 15, month 3, month 6
Vestibular function assessed at D15, M3 and M6 with: • presence or absence of a spontaneous and positional nystagmus • mean gains of the vestibulo-ocular reflex measured by the vHIT | At day 15, month 3, month 6

CONTACTS AND LOCATIONS:
Locations (1):
- Lariboisière Hospital, Paris, Île-de-France Region, France